CLINICAL TRIAL: NCT02438384
Title: Patient Education to Improve Pain Management in Older Adults With Acute Musculoskeletal Pain: A Pilot Randomized Trial
Acronym: BETTER_Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Federation for Aging Research (Other); The John A. Hartford Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0986
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-03

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Pts will receive education and follow-up based on judgment of emergency provider.
- Video (Experimental): Patients will watch 10 minute educational video
  Interventions: Behavioral: Video
- Video plus Phone Follow-up (Experimental): Patients will watch 10 minute educational video and receive phone call follow-up at 3 days to assess pain symptoms. Patients with a pain score of 4 or more will receive another call with advice from a geriatric pain specialist.
  Interventions: Behavioral: Video; Behavioral: Phone follow-up

INTERVENTIONS:
Behavioral: Video — This is a 10 minute interactive video which provided information to the viewer regarding the safe and effective use of analgesics for acute musculoskeletal pain at home. The focus is on acetaminophen, NSAIDs, and opioids.
  Arms: Video; Video plus Phone Follow-up
Behavioral: Phone follow-up — The call will be made by the study coordinator, who is a medical student. Any patients reporting a pain score in the past 24 hours of 4 or more will be re-contacted by an emergency physician with special training in geriatric pain management. This individual will provide recommendations to the patient regarding treatment options.
  Arms: Video plus Phone Follow-up

SUMMARY:
This is a three arm pilot randomized trial. Patients will be assigned to:

1. Usual care
2. Video education in the Emergency Department (ED)
3. Video education in the ED plus phone follow-up at three days with geriatric pain management specialist for all patients with pain >=4/10

DETAILED DESCRIPTION:
This is a three arm pilot randomized trial. Patients will be assigned to:

1. Usual care
2. Video education in the ED (10 minute interactive video)
3. Video education in the ED plus phone follow-up at three days with geriatric pain management specialist for all patients with pain >=4/10

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older; ED visit for acute musculoskeletal pain

Exclusion Criteria:

* Cognitively impaired; chronic pain (daily opioid use prior to onset of pain or pain symptoms more than one month); prison; injury or pain condition requiring hospital admission.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06-17 (Actual); Study Completion 2017-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Platts-Mills, MD, MSc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals Emergency Department, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Platts-Mills TF, Hollowell AG, Burke GF, Zimmerman S, Dayaa JA, Quigley BR, Bush M, Weinberger M, Weaver MA. Randomized controlled pilot study of an educational video plus telecare for the early outpatient management of musculoskeletal pain among older emergency department patients. Trials. 2018 Jan 5;19(1):10. doi: 10.1186/s13063-017-2403-8. PMID 29304831
- See also: Randomized controlled pilot study of an educational video plus telecare for the early outpatient management of musculoskeletal pain among older eme... - PubMed - NCBI — https://www.ncbi.nlm.nih.gov/pubmed/29304831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in an academic emergency department between September 2015 and March 2017 and the last participant was enrolled in March 2017. Due to unavailability of research assistants, the study was suspended during the winter of 2015 and 2017 and summer 2016.
Period: Overall Study
Arm/Group | Usual Care | Video | Video Plus Phone Follow-up
Started | 25 | 25 | 25
Completed | 17 | 19 | 21
Not Completed | 8 | 6 | 4
Not completed — Lost to Follow-up | 8 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Video | Video Plus Phone Follow-up | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (2.1) | 63 (2.1) | 61 (2.1) | 63 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 13 | 50
  Male | 7 | 6 | 12 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 19 | 17 | 56
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 8 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 25 | 75
Formal Education [Count of Participants; unit: Participants] — Categorized as: <High School, High School or General Educational Development, Some College, College Degree, or Post-Graduate Education Self-reported by patients
  Participants | 25 | 25 | 25 | 75
Home [Count of Participants; unit: Participants] — Categorized as: Private Home or Assisted Living or Nursing Home Self-reported by patients
  Participants
    Private Home | 24 | 25 | 25 | 74
    Assisted Living | 1 | 0 | 0 | 1
Daily Medications [Mean (Standard Deviation); unit: number of medications] — Self-reported by patients. Patients asked: How many different prescription medications do you take daily?
  number of medications | 4.8 (0.8) | 4.5 (0.8) | 4.2 (0.8) | 4.5 (0.8)
Self-Reported Health of Excellent, Very Good, or Good [Count of Participants; unit: Participants] — Patients were asked: In general, how do you rate your health? excellent, very good, good, fair, poor. Reported number of patients with excellent, very good, or good response. Population: data unavailable for one participant in usual care group n=24
  Patients self-reported health as good, very good or excellent; fair or poor
  Participants
    number analyzed (Participants) | 24 | 25 | 25 | 74
    (all) | 20 | 20 | 19 | 59
Chronic Musculoskeletal Pain [Count of Participants; unit: Participants] — Self-reported. Patients were asked: have you had daily pain in your bones, muscles, tendons, ligaments or joints (also known as musculoskeletal pain) for the past six months or longer?
  Participants | 11 | 13 | 11 | 35
Pain Due to Musculoskeletal Injury [Count of Participants; unit: Participants] — Self reported by patients. Patients were asked: Where is the pain that brought you into the emergency department located (abdomen, chest, head, skin, eye, ear, jaw, neck, chest (traumatic), shoulder, arm , back, hip, leg, other.
  Research assistant indicated if pain was musculoskeletal or not. Limb pain was excluded if it was known to be caused by a blood clot or ischemia.
  Participants | 10 | 12 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: Change in Pain from emergency department (ED) visit to 30 day follow-up phone call will be measured by calculating the difference between the maximum pain score in the ED and the patient reported average overall pain severity in the past week using the 0-10 numeric rating scale for both measures.Change in pain will be reported as a negative number if the pain decreases (i.e., 10 to 8 = -2). Higher scores indicate a worse outcome.
Time Frame: ED visit and 30 days post-ED visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Video | Video Plus Phone Follow-up
Number analyzed (Participants) | 17 | 19 | 21
score on a scale | -1.3 (2.9) | -2.4 (3.2) | -3.0 (2.6)
Statistical Analysis 1: Comparison: Usual Care vs Video Plus Phone Follow-up; Test type: Superiority; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [1.2 to 2.1]
Statistical Analysis 2: Comparison: Usual Care vs Video; Test type: Superiority; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.6 to 1.6]

2. Secondary Outcome: Number of Participants Experiencing Medication Side Effects
Description: Patients were asked if they experienced any of the following side effects: fatigue, drowsiness, trouble sleeping, trouble thinking, dizziness, unsteadiness, nausea, vomiting, constipation, abdominal pain, black or bloody stool, trouble urinating, loss of appetite, itching or shortness of breath. Patients were also queried about any other side effects they had that were not on the list.
  Participants reporting at least one side effect were included.
Time Frame: 30 days after ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Video | Video Plus Phone Follow-up
Number analyzed (Participants) | 17 | 19 | 21
Participants | 12 | 9 | 8

3. Secondary Outcome: Average Overall Pain at One Month
Description: Determined using 0-10 numerical rating scale to answer the question "What is the average amount of pain you have experienced over the last week on a scale of 0-10. where 0 means no pain and 10 means pain as severe as it could possibly be.
Time Frame: 30 days after ED visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Video | Video Plus Phone Follow-up
Number analyzed (Participants) | 17 | 19 | 21
score on a scale | 5.8 (2.8) | 4.9 (3.5) | 4.5 (2.9)

4. Secondary Outcome: Mean Physical Function Scores
Description: Using a measure of higher-level physical function based on walking, climbing stairs, and carrying bags - scores range from 0 to 12 with higher score indicating higher function.
Time Frame: 30 days after ED visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Video | Video Plus Phone Follow-up
Number analyzed (Participants) | 17 | 19 | 21
score on a scale | 2.8 (2.8) | 4.3 (4.0) | 5.2 (3.9)

ADVERSE EVENTS:
Time Frame: Beginning at the time of the emergency department visit and continuing through 30 days afterwards
Description: Medication side effects were not considered adverse events. Patients who reported 1 or more side effects received a call from the study physician per protocol procedures.
Arm/Group | Usual Care | Video | Video Plus Phone Follow-up
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT02438384/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT02438384/SAP_001.pdf